CLINICAL TRIAL: NCT06587867
Title: Efficacy, Safety and Tolerability of Efgartigimod in Patients with Seronegative Generalized Myasthenia Gravis: an Open-Label Study
Brief Title: Seronegative Myasthenia Gravis - Efgartigimod IV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Vera Bril, Principal Investigator, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN 001
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Efgartigimod; Generalized Myasthenia Gravis
Keywords: seronegative; generalized myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — efgartigimod alfa

STUDY DESIGN:
Intervention Model Description: open label administration of efgartigimod
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- efgartigimod (Other): active treatment with efgartigimod.
  Interventions: Biological: efgartigimod

INTERVENTIONS:
Biological: efgartigimod — active drug efgartigimod to be administer

SUMMARY:
This is to study the efficacy, safety and tolerability of efgartigimod in patients with seronegative generalized myasthenia gravis. This is an open label study. There will be 30 participants to enroll at University Health Network Toronto General Hospital. Study duration is 43 weeks from screening to end of study.

DETAILED DESCRIPTION:
There will be screening period that includes ECG, safety blood collection, collection of demographics, vital signs, questionnaires, weight, pregnancy test (if applicable), genetic test. If eligible, participants will have run-in period from week 2 to week 5. Baseline is at week 6. Induction phase will be weekly from week 7, 8, and 9. Maintenance phase will be once every 2 weeks thereafter. Observation period will have 4 visits, End of study is at week 43.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent document(s) indicating that the subject has been informed of all pertinent aspects of the trial. Subjects must be willing and able to comply with the protocol, complete study assessments, and return for follow-up visits.
* Male or female subjects ≥ 18 years old.
* Diagnosis of SN MG defined as: (a) clinical syndrome consistent with a diagnosis of MG, and not otherwise explained by another condition, (b) abnormal neuromuscular transmission test results demonstrated by single-fiber electromyography or repetitive nerve stimulation; and (c) negative serologic test for anti-AChR and anti- MuSK antibodies as confirmed at screening, (d) limited, if any, response to therapy with immunotherapy and/or antiacetylcholinesterase (AChE) treatment. Further testing for low affinity antibodies to rapsyn-clustered AChR by cell-based assays will be done at baseline and the results included as part of subgroup analysis. All patients will have a negative genetic test for congenital myasthenic syndromes by history or at baseline to exclude the possibility of congenital myasthenic syndrome mimicking SN MG.
* MGFA Clinical Classification Class II, III, or IV at the time of screening and baseline.
* Moderate to severe myasthenia gravis as defined by a generalized myasthenia gravis impairment index score > 11 or MG-ADL score of at least 5 (with >50% of the score due to non-ocular symptoms) and a PASS response of "No" and a SSQ of < 70% with at least 6 months of historical data as the baseline.
* Stable or worsening MG as defined by MGII remaining stable or increasing in the 4 week run-in interval.
* Patients are required to be on a stable dose of their MG treatment (Standard of care-SoC) for at least one month prior to screening. The SoC is limited to AChE inhibitors, steroids and NSISTs (e.g., azathioprine, methotrexate, cyclosporine, tacrolimus, and mycophenolate mofetil. There is no requirement for specific generalised myasthenia gravis therapies.
* Patients who discontinued early from previous trials of efgartigimod for reasons other than pregnancy, rescue therapy or a SAE can be included.
* Females of childbearing potential who are sexually active with a non-sterilized male partner must be willing to use at least one highly effective contraception method from the time of screening and for 3 months after the final dose of efgartigimod.
* Non-sterilized males who are sexually active with a female partner of childbearing potential must be willing to use a condom for the duration of the study and for 3 months after the last dose of efgartigimod. Because male condom is not a highly effective contraception method, it is strongly recommended that female partners of a male study subject also use a highly effective method of contraception throughout this period.
* Vital signs, electrocardiogram (ECG), and laboratory parameters within the normal ranges at screening, or, if outside normal ranges, deemed not clinically significant by the Investigator.
* Patient has documented IgG >6 g/L within one month of screening
* Vaccinated for COVID-19 at least 2 weeks prior to screening visit.

Exclusion Criteria:

* Patients who discontinued early from trials of efgartigimod for pregnancy or rescue reasons or an SAE that was likely to result in a life-threatening situation or pose a serious safety risk.
* Pregnant and lactating women, and those intending to become pregnant during the trial or within 3 months after the last dosing. Women of childbearing potential should have a negative urine pregnancy test at screening and baseline.
* Male patients who are sexually active and do not intend to use effective methods of contraception (as mentioned above) during the trial or within 3 months after the last dosing or male patients who plan to donate sperm during the trial or within 3 months after the last dosing.
* Patients with known hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) seropositivity.
* Patients with known autoimmune disease other than MG (e.g., rheumatoid arthritis) which in the investigator opinion would interfere with an accurate assessment of clinical symptoms.
* Patients with clinical evidence of other significant disease or patients who underwent a recent major surgery, which could confound the results of the trial or put the patient at undue risk.
* Patients with renal/hepatic function impairment as defined by (Cr>1.5 x elevated) and/or (transaminases > 2.5 x elevation) at screening.
* Patients with known medical history of hypersensitivity to any of the ingredients of efgartigimod.
* Patients who have received rituximab or eculizumab in the 6 months before screening.
* Patients who have undergone thymectomy within 3 months of screening.
* Patients who had intravenous immunoglobulin or plasma exchange within 4 weeks of screening.
* Patient who has clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection at screening
* Patient has received a live or a live-attenuated vaccination during the month before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Total Myasthenia Gravis Impairment Index (MGII) score | through study completion for 42 weeks
  Myasthenia Gravis Impairment Index (MGII) is a composite score based on a patient self-reported multidomain questionnaire as well as physician-documented clinical measures. MGII has 22 patient-reported and 6 physician-assessed items with a final composite score of 84, with higher score signifying greater disability.

SECONDARY OUTCOMES:
MG-ADL (Myasthenia Gravis-Activities of Daily Living) | through study completion for 42 weeks
  The MG-ADL is an 8-item patient-reported scale to assess MG symptoms and their effects on daily activities. The MG-ADL total score range is 0-24, with higher scores indicative of greater disease severity.
QMG (Quantitative Myasthenia Gravis) score | through study completion for 42 weeks
  The QMG scale quantifies disease severity based on impairments of body functions and structures as defined by the International Classification of Disability and Health. The QMG scale consists of 13 items that measure endurance or fatigability, and accounts for fluctuations in disease state. The QMG total score range is 0-39, with higher scores indicative of greater disease severity.
MG-QOL (Myasthenia Gravis Quality of Life) | through study completion for 42 weeks
  MG-QOL revised consists of 15 items/ question. These include mobility (9 items), symptoms (3 items), and contentment and emotional well-being (3 items). Items are scored in a Likert scale from 0 to 4 and the total sum score ranges from 0 to 60, where higher scores indicate worse HRQoL.
PASS (Patient Acceptable Symptom State) response | through study completion for 42 weeks
  The PASS response is based on a dichotomous 'Yes' or 'No' response, asking whether a patient is satisfied overall with their current status and thus measures holistic satisfaction with their MG state. The PASS response of "Yes" has been shown to correlate with a favourable MGII and the simple single question (SSQ, percentage of normal).
Single Simple Question (SSQ) | through study completion for 42 weeks
  The SSQ is a question that asks what percentage of normal that the patient feels with respect to their MG. A SSQ threshold ≥72.5% out of normal at 100% predicts an acceptable MG state.
Myasthenia Gravis Foundation of America (MGFA) | through study completion for 42 weeks
  The MGFA classes are pure ocular (class I), mild generalized (class II), moderate generalized (class III), severe generalized (class IV), and intubation/myasthenic crisis (class V). Within the generalized categories II, III, and IV, patients are subclassified as class A if their symptoms are predominantly generalized or class B if their symptoms are predominantly bulbar. The MGFA also has a system to classify patients based on postintervention outcomes and includes remission, defined as 1 year or longer without signs or symptoms and without any symptomatic (pyridostigmine) treatment, and which can be divided in complete (no pharmacologic treatment at all) or pharmacologic remission. Minimal manifestation status is defined as minimal signs or symptoms (no specific timeframe was defined) and pyridostigmine use may be accepted.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Bril, MD, Principal Investigator — Toronto General Hospital
Locations (1):
- University Health Network, Division of Neurology, Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Khateb M, Sivadasan A, Barnett-Tapia C, Daniyal L, Fernando L, Chen S, Lovblom LE, Katzberg H, Bril V. Open-label study of efgartigimod in seronegative myasthenia gravis. Ther Adv Neurol Disord. 2025 Oct 31;18:17562864251388019. doi: 10.1177/17562864251388019. eCollection 2025. PMID 41180124